CLINICAL TRIAL: NCT05130502
Title: Investigation of the Effect of Foam Roller and Kinesiotape Application on Performance Parameters, Pain and Fatigue
Brief Title: Investigation of the Effect of Foam Roller and Kinesiotape Application on Performance Parameters, Pain and Fatigue With Football Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Pamukkale University (Other)
Collaborators: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Muhammet Alper Karabag, Physiotherapist, Master Degree student, Pamukkale University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: MAKarabag
Record Dates: First submitted 2021-10-28; First posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Performance; Pain; Fatigue
Keywords: Foam roller; Kinesiotaping; Dynamic warm up; Performance
MeSH Terms: conditions — Pain; Fatigue | interventions — Athletic Tape

STUDY DESIGN:
Intervention Model Description: Individuals will perform foam roller and dynamic warm up and kinesiotape and dynamic warm up. there will be one week wash-out between tests.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foam roller (Experimental): Individuals perform Foam roller on bilateral legs and the muscles include Quadriceps, hamstring and gastrocnemius and soleus with a dynamic warm up program The investigators conduct the test for 2 sets and 60 seconds with 30 seconds rest period per muscle
  Interventions: Other: Foam roller
- Kinesiotape (Active Comparator): Individuals perform Kinesiotape on bilateral legs and the muscles include Quadriceps, hamstring and gastrocnemius and soleus with a dynamic warm up program The investigators conduct the kinesiotape per muscle and will wait for 45 minutes for bring out the effects.
  Interventions: Other: Kinesiotape

INTERVENTIONS:
Other: Foam roller — The investigators use Foam roller to 3 muscle groups per leg then conduct a dynamic warm up program and conduct performance tests
  Arms: Foam roller
Other: Kinesiotape — The investigators use Kinesiotape to 3 muscle groups per leg, wait 45 minutes for bring out the effects then conduct a dynamic warm up program and conduct performance tests
  Arms: Kinesiotape

SUMMARY:
The aim of our study is to compare the effects of foam roller plus dynamic stretching and kinesiotape plus dynamic stretching on performance parameters,pain and fatigue in football players. The results of our study will show the effects of the best choice between applications and help to reduce waste of time.

DETAILED DESCRIPTION:
The aim of our study is to compare the effects of foam roller plus dynamic stretching and kinesiotape plus dynamic stretching on performance parameters,pain and fatigue in football players. The results of our study will show the effects of the best choice between applications and help to reduce waste of time. Performance parameters include; flexibility, dynamic reaction time, sprint and agility.

The hypotheses the investigators will test for this purpose; H1: Foam Roller application is more effective on performance parameters than Kinesiotape application. H2: Foam Roller application is more effective on pain than Kinesiotape application. H3: Foam Roller application is more effective on fatigue than Kinesiotape application.

ELIGIBILITY:
Inclusion Criteria:

* Playing in Aydın Adnan Menderes University Football Team and volunteering.

Exclusion Criteria:

* Individuals with medical conditions that may affect their ability to complete the work, such as recurrent muscle, bone, tendon, and ligament injuries, or a history of prior lower extremity surgery.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-11-21 (Estimated); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
Muscle Pain | immediately after application
  With VAS scale ; The scale goes from '0' to '10' points. A score of 0 means 'I have no pain' and a score of 10 means 'I have very severe pain'.
Fatigue | immediately after application
  With BORG scale; The scale goes from '0' to '10' points. 0 points means 'I am not tired at all' and 10 points means 'I have very severe fatigue'.
Sprint | in 1 hour after application
  20m sprint test; 20-meter sprint test will be applied in the study. Participants will be positioned with one foot in front of the other and not crossing the starting line. Swinging movements to the right-left or forward-backward will not be allowed before the run. Participants will run a single max sprint at 20 meters and sprint time will be recorded using an automatic light switch system (SMARTSPEED™, Fusion Sport Inc., Australia; 1000 Hz). A single measurement will be taken from subjects
Agility | in 1 hour after application
  The 18.3 m pro-agility (505) test will be applied. The test will start from 3 pontoons that are 4.6 meters from each other, over the middle pontoon. The individual will run 4.6 m to the pontoon on the left first. After his foot contacts the line (followed by the line judge), he will turn around and run up to the pontoon located 9.1 m to the right (4.6 m to the right of the center line) and again to touch the line with his foot. After making contact with the right line, it will turn and run towards the center pontoon. The best time of two attempts will be recorded as agility speed. Participants will rest for 1 minute between trials. All measurements will be performed using (Fusionsports Smartspeed™ PRO photocell, Fusion Sport, Queensland, Australia).
Dynamic reaction time | in 1 hour after application
  Dynamic reaction time (DRT) will be evaluated using the Blazepod system, which includes "pods" equipped with touch sensors and LED lights. Three of the blazepod pods will be affixed to a wall 1.5 m above the floor, each 1.5 m apart. During testing, when a random single bin is lit, the subject will be instructed to react as quickly as possible by running towards the light and touching the bin. Subjects will do so with a total of 6 randomized light triggers for a single trial. Subjects will perform 2 trials with 3 minutes rest. Average reaction time will be calculated for each trial and the best score will be used for analysis.
Flexibility | in 1 hour after application
  The investigators use 'Hudl' tecnique. Hip and knee flexion measurements will be calculated with digital goniometer in supine (for hip) and prone (for knee) positions. 3 trial will be taken and will be averaged. With the Hudl technique, the necessary angles will be measured with the help of the smartphone.

CONTACTS AND LOCATIONS:
Locations (1):
- Aydın Adnan Menderes University, Aydin, Efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No